CLINICAL TRIAL: NCT06824103
Title: A Single-arm Multi-center Study of Ruxolitinib in Chinese Participants With Corticosteroid-refractory Chronic Graft Versus Host Disease After Allogeneic Stem Cell Transplantation
Brief Title: Study of Efficacy and Safety of Ruxolitinib in Chinese Participants With Corticosteroid-refractory Chronic Graft vs. Host Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424D2413
Record Dates: First submitted 2025-02-04; First posted 2025-02-13 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Graft vs. Host Disease; Chronic Graft vs. Host Disease; Corticosteroid-refractory Chronic Graft vs. Host Disease
Keywords: cGvHD; GvHD; SR-cGvHD; ruxolitinib; INC424; Chinese adult; Pediatric; Corticosteroid; refractory
MeSH Terms: conditions — Graft vs Host Disease | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): Chinese participants (adult and pediatric) who will receive ruxolitinib daily.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib is taken orally daily at 10 mg BID, given as two 5 mg tablets.
  Other Names: INC424

SUMMARY:
The purpose of the study is to assess the efficacy and safety of ruxolitinib in Chinese adult and pediatric participants aged 12 years or older with corticosteroid-refractory chronic graft vs. host disease (SR-cGvHD).

DETAILED DESCRIPTION:
This is a single arm, multi-center, open label study which will enroll approximately 50 participants and investigate the efficacy and safety of ruxolitinib administered in adult and adolescent (≥12 years old) Chinese participants with SR-cGvHD.

The total duration on study for an individual participant will be up to 164 weeks (approximately 3 years).

The study consists of following periods, with each cycle comprised of 4 weeks (28 days):

* Screening Period (Day -28 to Day -1)
* Treatment period (Day 1 to Cycle 39/EOT)
* Safety follow-up (Last dose +30 days)
* Long-term survival follow-up period (EOT to 156 weeks on study).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Male or female Chinese participants aged 12 or older at the time of informed consent
* Able to swallow tablets.- Have undergone alloSCT from any donor source (matched unrelated donor, sibling, haplo-identical) using bone marrow, peripheral blood stem cells, or cord blood. Recipients of non-myeloablative, myeloablative, and reduced intensity conditioning are eligible.
* Evident myeloid and platelet engraftment:

  * Absolute neutrophil count (ANC) >1,000/mm3 AND
  * Platelet count ≥25,000/mm3

Note: Use of growth factor supplementation and transfusion support is allowed during the trial, however, transfusion to reach a minimum platelet count for inclusion is not allowed during screening and at baseline.

* Participants with clinically diagnosed cGvHD staging of moderate to severe according to NIH Consensus Criteria (Jagasia et al 2015) prior to Cycle 1 Day 1.

  * Moderate cGvHD: at least one organ (not lung) with a score of 2, 3 or more organs involved with a score of 1 in each organ, or lung score of 1.
  * Severe cGvHD: at least 1 organ with a score of 3, or lung score of 2 or 3.
* Participants currently receiving systemic corticosteroids for the treatment of cGvHD for a duration of < 12 months prior to Cycle 1 Day 1, and have a confirmed diagnosis of corticosteroid refractory cGvHD defined per 2014 NIH consensus criteria (Martin et al 2015) irrespective of the concomitant use of a calcineurin inhibitor, as follows:

  * A lack of response or disease progression after administration of minimum prednisone 1 mg/kg/day for at least 1 week (or equivalent) OR
  * Disease persistence without improvement despite continued treatment with prednisone at >0.5 mg/kg/day or 1 mg/kg/every other day for at least 4 weeks (or equivalent) OR
  * Increase to prednisone dose to >0.25 mg/kg/day after two unsuccessful attempts to taper the dose (or equivalent)
* Participants has Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria:

For a full list of exclusion criteria, refer to Section 5.2. Key exclusion criteria include

* Participants who have received two or more systemic treatments for cGvHD in addition to corticosteroids ± CNI for cGvHD.
* Participants who have received ROCK2 inhibitors for cGvHD.
* Participants that transition from active aGvHD to cGvHD without tapering off corticosteroids ± CNI and any systemic treatment

Note: Participants receiving up to 30 mg by mouth once a day of hydrocortisone (i.e., physiologic replacement dose) of corticosteroids are allowed.

* Participants who were treated with prior JAK inhibitors for aGvHD; except when the participant achieved complete or partial response and has been off JAK inhibitor treatment for at least 8 weeks prior to Cycle 1 Day 1.
* Failed prior alloSCT within the past 6 months from Cycle 1 Day 1.
* Participants with relapsed primary malignancy, or who have been treated for relapse after the alloSCT was performed.
* SR-cGvHD occurring after a non-scheduled donor lymphocyte infusion (DLI) administered for pre-emptive treatment of malignancy recurrence. Participants who have received a scheduled DLI as part of their transplant procedure and not for management of malignancy relapse are eligible.

Other protocol-defined inclusion/exclusion may apply.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2029-11-29 (Estimated); Study Completion 2032-01-11 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Cycle 7 Day 1; each Cycle =28 days
  ORR is defined as the percentage of participants demonstrating a complete response (CR) or partial response (PR) without the requirement of additional systemic therapies for an earlier progression, mixed response or non-response, according to National Institute of Health (NIH) Consensus Criteria.

SECONDARY OUTCOMES:
Failure-free Survival (FFS) | up to 3 years
  FFS is defined as the time from the date of start of study treatment to the earliest of: i) relapse or recurrence of underlying disease or death due to underlying disease, ii) nonrelapse mortality, or iii) addition or initiation of another systemic therapy for cGvHD.
Best Overall Response (BOR) | at any point up to cycle 7 day 1 (each cycle is 28 days) or the start of additional systemic therapy for cGvHD, approx. 6 months
  Percentage of participants who achieved overall response (CR+PR) at any time point (up Cycle 7 Day 1 or the start of additional systemic therapy for cGvHD).
ORR at end of cycle 3 | end of cycle 3; each cycle = 28 days
  Percentage of participants who achieved overall response (CR+PR) at Cycle 4 Day 1.
Duration of Response (DOR) | from first response until cGvHD progression, death, or the date of addition of systemic therapies for cGvHD, approx.36 months
  DOR is assessed for responders only and is defined as the time from first response until cGvHD progression, death, or the date of addition of systemic therapies for cGvHD.
Overall Response (OS) | from the date of study treatment (ruxolitinib) initiation to the date of death due to any cause, approx. 36 months
  OS is defined as the time from the date of study treatment (ruxolitinib) initiation to the date of death due to any cause.
Non-Relapse Mortality (NRM) | from date of study treatment (ruxolitinib) initiation to date of death not preceded by underlying disease relapse/recurrence, approx. 36 months
  NRM is defined as the time from date of study treatment (ruxolitinib) initiation to date of death not preceded by underlying disease relapse/recurrence.
Malignancy Relapse/Recurrence (MR) | from date of study treatment to hematologic malignancy relapse/recurrence, approx. 36 months
  Malignancy relapse/recurrence is defined as the time from date of study treatment to hematologic malignancy relapse/recurrence.
Reduction of daily corticosteroids dose at cycle 7 day 1 | Cycle 7 Day 1; each cycle = 28 days
  Systemic corticosteroid use is the percentage of participants with >=50% reduction from baseline in daily corticosteroid dose, the proportion of subjects with reduction from baseline to ≤ 0.2 mg/kg/day methylprednisolone (or equivalent dose of ≤ 0.25 g/kg/day prednisone or prednisolone), and subjects successfully tapered off all systemic corticosteroids at Cycle 7 Day 1, by time intervals and overall.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- China (17):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Guiyang, Guizhou
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Ningbo, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Changsha
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Shanhecun

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com